CLINICAL TRIAL: NCT04338113
Title: EARLY-MYO-Myocarditis (EARLY Assessment of MYOcardial Tissue Characteristics by CMR in Myocarditis) Registry
Brief Title: EARLY-MYO-Myocarditis Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-MYO-Myocarditis
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to depict the myocardial tissue characteristics in patients with myocarditis by CMR and other cardiac imaging modalities and to assess the prognostic value of imaging-derived indices. Information will be collected prospectively in about 200 patients with myocarditis in 5 sites. Subjects will be followed for up to 5 years.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational registry study of patients with myocarditis that undergo CMR examination. Information of other cardiac imagings and clinical outcomes are also prospectively collected in the database. This project will establish a prospective registry of 200 patients with myocarditis in 5 sites with follow-ups of up to 5 years.

The aim of the project will be as following:

1. To investigate myocardial tissue features and functional changes in patients with myocarditis.
2. To identify CMR-derived indices that are associated with adverse clinical outcomes.
3. To compare CMR with other alternative cardiac imaging modalities (i.e., echocardiography or SPECT) on prognostic prediction in patients with myocarditis.

ELIGIBILITY:
[Inclusion Criteria]:

1. Definitive diagnosis of myocarditis - A definitive diagnosis of myocarditis is based upon identification of diagnostic findings on EMB, including histology (Dallas criteria) as well as immunohistochemical stains.
2. Criteria for clinically suspected myocarditis - We adopted the 2013 European Society of Cardiology (ESC) position statement criteria for "clinically suspected" myocarditis, which require that a patient have at least one of the following clinical presentations of myocarditis and at least one diagnostic criteria; if the patient is asymptomatic at least two diagnostic criteria are required. A diagnosis of clinically suspected myocarditis also generally requires the absence of other clinical conditions that could explain the clinical findings such as cardiovascular disease (eg, angiographically significant CAD [coronary stenosis ≥50%], valve disease, or congenital heart disease), or an extra-cardiac condition (eg, hyperthyroidism). While it is possible to make a diagnosis of "clinically suspected" myocarditis in a patient with a concomitant condition such as CAD, clinical findings must be carefully reviewed to determine whether findings can be explained by a single disease process or whether the patient likely has at least two separate conditions. Clinical suspicion is higher with greater numbers of fulfilled criteria unrelated to other conditions .

   * Clinical presentations:

     * Acute chest pain (pericarditis or pseudo-ischemic)
     * New-onset (days up to three months) or worsening of dyspnea at rest or exercise, and/or fatigue, with or without left and/or right HF signs
     * Palpitation, and/or unexplained arrhythmia symptoms and/or syncope, and/or aborted sudden cardiac death
     * Unexplained cardiogenic shock
   * Diagnostic criteria:

     * ECG/Holter stress test features - New 12-lead ECG and/or Holter and/or stress testing abnormalities with any of the following: first to third degree atrioventricular (AV) block or bundle branch block, ST/T wave change (ST elevation or T wave inversion), sinus arrest, ventricular tachycardia or fibrillation, asystole, atrial fibrillation, significantly reduced R wave height, intraventricular conduction delay (widened QRS complex), abnormal Q waves, low voltage, frequent premature beats, or supraventricular tachycardia.
     * Elevated troponin T or troponin I.
     * Functional and structural abnormalities on cardiac imaging (echocardiogram, angiogram, or CMR) - New, otherwise unexplained abnormality of LV and/or RV function (regional wall motion abnormality or global systolic or diastolic dysfunction); such abnormality may occur with or without one or more of the following: ventricular dilatation, increased ventricular wall thickness, pericardial effusion or intracavitary thrombus.
     * Tissue characterization by CMR - Late gadolinium enhancement (LGE) and/or findings consistent with edema in pattern suggestive of myocarditis. (See 'Cardiovascular magnetic resonance' below.)
   * The following ancillary features support the clinical suspicion of myocarditis:

     * Fever ≥38.0 degrees C at presentation or during the preceding 30 days with our without associated symptoms (eg, chills, headache, myalgias, malaise, decreased appetite, nausea, vomiting, or diarrhea).
     * Prior clinical suspected or definite myocarditis.
     * Exposure to toxic agents.
     * Extra-cardiac autoimmune disease.

[Exclusion Criteria]:

1. Patient who is unable to comply with the follow-up schedule.
2. Patient who has any medical conditions that in the opinion of the investigators will not be appropriate to participate in the study.
3. Patient has a life expectancy of less than 6 months due to any condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with myocarditis undergo CMR examination are eligible for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcomes of adverse cardiac events | 1 year
  cardiac death，sudden deatch, malignant arrhythmias，heart failure and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China